CLINICAL TRIAL: NCT00726440
Title: Are the Continous Glucose Monitoring Systems Able to Improve Long Term Glycaemic Control in Type 1 Diabetic Patients With Poor Metabolic Control?
Brief Title: Are the Continuous Glucose Monitoring Systems Able to Improve Long Term Glycaemic Control in Type 1 Diabetic Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-A01022-51
Record Dates: First submitted 2008-07-23; First posted 2008-08-01 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2011-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Real Time Continuous Glucose Monitoring System; HbA1c; Navigator®
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group1-patient (Active Comparator): The patient will be encouraged to use the Navigator® all the time and to modify his treatment according to the continous blood glucose measurements. The patients will follow an educational process in order to adapt insulin doses according to each sensor data.
  Interventions: Device: Navigator®
- Group2-diabetologist (Active Comparator): The patient will follow the same educational process as group 1 concerning insulin dose adaptation. They will use the continous glucose monitoring device according to the diabetologist's prescription and they will receive precise instructions to make considering results. The duration of the use of the Navigator® will be increased if one of the following criteria is observed at the consultation each 3 months:
  * HbA1c>=7.5%
  * 1 severe hypoglycaemia or more
  * More than 4 benign hypoglycaemia per week
  According to these criteria, every 3 months, the duration of the use of the monitoring system will be increased as following:
  * step 1: 3 sensors per month
  * step 2: 4 sensors per month
  * step 3: 5 sensors per month
  * step 4: continuous use
  Interventions: Device: Navigator®
- Group3-Control (Placebo Comparator): Usual follow up with self-monitoring blood glucose.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Navigator® — Patients will be encouraged to use the Navigator® all the time and to modify their treatment according to the device measurments. Patients will also follow and educational process in order to adapt insulin doses according to each sensor data
  Arms: Group1-patient
Device: Navigator® — Patients will follow the same educational process as group1 concerning insulin doses adaptation.The duration of the use of the devicewill be determined at the consultation every each 3 months.
  Arms: Group2-diabetologist
Device: Placebo — Patients will have their usual follow up with self-monitoring blood glucose
  Arms: Group3-Control

SUMMARY:
The "Capteur Evadiac" study group, composed of French and Belgian diabetologists, has designed a 1 year randomized controlled multicenter study in order to define what should be the best clinical way of using continuous glucose monitoring in the long term to improve metabolic control in uncontrolled type 1 diabetes patients.

DETAILED DESCRIPTION:
The primary objective of the study is to determine whether patients with chronically poor glycaemic control as evidenced by HbA1c >= 8% twice can achieve improved metabolic control using during one year CGM together with educative program about insulin adaptation doses compared to conventional self monitoring finger sticks with educative program about insulin adaptation doses alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes for ≥ 12 months or more (including Cpeptide negative secondary diabetes)
* Children between 8 and 18 years old
* Adults between 18 and 60 years old
* Patients treated with basal-bolus insulin regimens, pump or multiple daily injection, only with analogs, for at least 6 months
* Performing at least 2 finger sticks glucose controls per day
* Able and motivated to use the device
* HbA1c ≥ 8% twice with HPLC method(DCA 2000 excluded)
* Written informed consent obtained prior to enrollment in the study

Exclusion Criteria:

* Blindness or impaired vision so the screen cannot be recognized
* Allergy to sensor
* Active proliferative retinopathy not stabilized by laser or vitrectomy occurence in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgical treatment during study
* Treatment with systemic corticosteroid or medication known to influence insulin sensitivity in the 3 months prioir to visit 1
* Pregnancy
* Manifest psychiatric disturbance
* Presence of any conditions (medical, including clinically significant abnormal laboratory test, psychological, social or geographical) actuel or anticipated that the investigators feels would compromise the patient safety or limit his/her successful participation in the study.
* Hemoglobinopathy that interfers with HbA1c measurement

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Comparison of HbA1c mean between the 3 groups | at 1 year

SECONDARY OUTCOMES:
Comparison of glucose stability in the 3 groups | inclusion, M3, M6, M9, M12
Frequency of severe hypoglycaemic episodes and ketoacidosis episodes during the study period | study period
Frequency of symptomatic benign hypoglycaemic episodes during the week prior to each visit. inclusion and prior to M3, M6, M9, M12 | prior to inclusion and prior to M3, M6, M9, M12
Comparison of HbA1c in patients treated by pump to those treated by multiple daily injection | inclusion, M3, M6, M9, M12
Evaluation of the Quality of Life (DQOL and SF36) and patient's satisfaction in the 3 groups | inclusion and M12
Comparison of weight, insulin doses, in each group | study period
comparison of the sensors consumption in group 1 and 2 and the evolution in time of this consumption | study period

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Riveline, MD, Study Director — CH Sud Francilien
Locations (19):
- CHU Sart Tilman Liège, Liège, Belgium
- France (18):
  - CHU Jean Minjoz, Besançon, Besancon
  - CH SUD Francilien, Corbeil-Essonnes, Corbeil Essonnes
  - University Hospital Grenoble, Grenoble, Grenoble
  - Hopital Edouard Herriot, Lyon, Lyon
  - CHU Marseille Hôpitaux Sud, Marseille, Marseille
  - Chu Montpellier, Montpellier, Montpellier
  - CHU Hôpital Jeanne d'Arc, Nancy, Nancy
  - CHU Nantes, Nantes, Nantes
  - Hopital Hotel Dieu, Paris, Paris
  - Hopital Haut Leveque, Pessac, Pessac
  - CHU Rennes, Rennes, Rennes
  - Hopital Bellevue, Saint-Etienne, Saint Etienne
  - CHU Toulouse, Toulouse, Toulouse
  - CHU La Pitié Salpetrière, Paris
  - CHU Robert Debré, Paris
  - CHU de Reims-Hôpital Américain, Reims
  - CHU de Reims-Hôpital Robert debré, Reims
  - CHU Strasbourg, Strasbourg

REFERENCES:
- [Derived] Riveline JP, Schaepelynck P, Chaillous L, Renard E, Sola-Gazagnes A, Penfornis A, Tubiana-Rufi N, Sulmont V, Catargi B, Lukas C, Radermecker RP, Thivolet C, Moreau F, Benhamou PY, Guerci B, Leguerrier AM, Millot L, Sachon C, Charpentier G, Hanaire H; EVADIAC Sensor Study Group. Assessment of patient-led or physician-driven continuous glucose monitoring in patients with poorly controlled type 1 diabetes using basal-bolus insulin regimens: a 1-year multicenter study. Diabetes Care. 2012 May;35(5):965-71. doi: 10.2337/dc11-2021. Epub 2012 Mar 28. PMID 22456864